CLINICAL TRIAL: NCT06381739
Title: A Phase 2 Trial to Evaluate Safety and Immunogenicity of a Next-generation COVID-19 Vaccine Delivered by Inhaled Aerosol to Humans
Brief Title: A Trial of a Next Generation COVID-19 Vaccine Delivered by Inhaled Aerosol
Acronym: AeroVax
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M011
Record Dates: First submitted 2024-04-23; First posted 2024-04-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChAd-triCoV/Mac (Experimental): ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- Control (Placebo Comparator): Placebo
  Interventions: Other: Control

INTERVENTIONS:
Biological: ChAd-triCoV/Mac — Clinical-grade, fully certified ChAd-triCoV/Mac produced according to current Good Manufacturing Principles (cGMP) will be provided. A single dose of ChAd-triCoV/Mac diluted in 0.5mL formulated buffer will be aerosolized and inhaled via a mouthpiece and tidal breathing over approximately 2 minutes using the AeroNeb Solo Mesh Nebulizer.
  Arms: ChAd-triCoV/Mac
Other: Control — A single dose of placebo (0.5mL formulated buffer) will be aerosolized and inhaled as the intervention vaccine.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to study the safety of a new inhaled vaccine to prevent COVID infection and learn about the immune responses that are made in the lungs and the blood after vaccination. Participants will be randomized (like the toss of a coin) to receive the experimental vaccine or a placebo (a look-alike solution that contains no vaccine).

To be in the study participants will have to have already had three doses of a messenger ribonucleic acid (mRNA) COVID vaccine and be generally healthy. Participants are given a single dose of the vaccine by breathing in a fine mist that goes directly into the lungs.

During follow-up participants will:

* visit the clinic for checkups and blood tests at 2, 4 and 8 weeks after vaccination
* report their symptoms for 24 weeks after getting the vaccine.

In some participants, the researchers will collect cells from the lung 4 weeks after vaccination (a test known as a bronchoscopy).

DETAILED DESCRIPTION:
The global impact of the coronavirus disease 2019 (COVID-19) pandemic remains profound; COVID-19 continues to be one of the leading causes of death and hospitalization due to infectious disease, disproportionately affecting the elderly and immunocompromised. The continuous evolution of the virus has significantly challenged the effectiveness of first-generation and updated vaccination strategies. These variants of concern (VOCs) can evade neutralizing antibodies.

Adequate and early lung mucosal immunity is critical for control of infection but current vaccines fail to induce robust mucosal immunity in the lungs, a major reason for the high rates of break-through infections. The respiratory mucosal route of immunization, however, can induce protective respiratory mucosal immunity consisting of trained innate immunity (via memory airway macrophages), mucosal antibodies, and tissue-resident memory CD4+/CD8+ T cells.

A phase 1 study has been completed using a recombinant chimpanzee adenovirus (ChAd) vector, ChAd-CoV3/Mac in 23 healthy volunteers and has shown that the vaccine can be safely administered by aerosol and that immune responses against COVID-19 develop in the lung and T-cells and neutralizing antibodies are generated in the blood.

The purpose of this placebo-controlled Phase 2 trial is to determine if this new COVID-19 vaccine, ChAd-triCoV/Mac, is safe to give by aerosol to people who have been vaccinated with at least three doses of a COVID mRNA vaccine and evaluate the immune responses generated. Specifically, the researchers want to see if T cell responses and antibody responses to the COVID virus proteins develop in the blood after receiving the vaccine.

There is a lack of surrogate immune markers for vaccine-induced protection against antibody-evading VOCs of SARS-CoV-2. However, given the now recognized importance of respiratory mucosal T cell immunity in anti-SARS-CoV-2 host defense, this study will allow for a correlation of mucosal T cell immunity with the T cells in blood to help predict vaccine efficacy, and inform the design of phase 3 efficacy studies.

ELIGIBILITY:
Inclusion criteria:

1. Adults who are 18-65 years old on the day of randomization (day 1)
2. Able to read, write and communicate using the English or French language.
3. Received at least 3 doses of an mRNA COVID vaccine.
4. Individuals of childbearing potential must have a negative pregnancy test prior to vaccination and be willing to practice effective contraception for 8 weeks post-vaccination.
5. Able to understand and comply with protocol requirements and instructions; able to report adverse events; able to attend scheduled study visits and complete required investigations.
6. For participants in the BAL sub-study, Complete Blood Count (CBC) and chemistry (creatinine) within normal limits.
7. For participants in the BAL sub-study, forced expiratory volume in 1 second (FEV1) > the lower limit of normal (LLN), and FEV1/FVC (forced expiratory volume in 1 second/forced vital capacity) ratio above the LLN.
8. Agree not to enroll in any other intervention studies for the duration of the study where the intervention could be reasonably expected to be associated with adverse events overlapping with the inhaled vaccine or the immune responses being measured.

Exclusion criteria:

1. Failure to provide informed consent.
2. Women who are pregnant or breastfeeding.
3. Have received any recombinant adenoviral-vectored COVID-19 vaccine (AstraZeneca [Vaxzeria] or Johnson & Johnson (Janssen Jcovden).
4. COVID infection (positive PCR or antigen (Ag) test, self-reported or lab documented) within the last 90 days.
5. Last dose of a COVID vaccine administered less than 90 days prior to study entry.
6. Administration of any vaccine within 2 weeks of study entry.
7. Active pulmonary disease diagnosed by a physician including asthma, chronic bronchitis, interstitial lung disease, pulmonary hypertension, lung cancer, cystic fibrosis, or bronchiectasis. Current use of daily inhaled steroids for any condition.
8. Persons with HIV and a detectable HIV viral load (>20 copies/mL), self-reported or confirmed.
9. Administration of monoclonal antibodies for treatment of COVID-19 infection within 3 months.
10. Moderately or severely immunocompromised (e.g. transplant recipients/CAR-T cell therapy, currently on chemotherapy for cancer or on potent immunosuppressant therapies e.g. rituximab or high dose steroids [>30 mg of prednisone equivalent daily], or moderate or severe primary immunodeficiency syndrome).
11. History of severe reaction to previous COVID vaccination (e.g. hives, difficulty breathing, high fever, seizures, myocarditis, pericarditis)).
12. Potential contraindication to COVID vaccination (e.g. venous or arterial thrombosis with thrombocytopenia after vaccination, history of cerebral venous thrombosis with thrombocytopenia, history of heparin induced thrombocytopenia, history of myocarditis or pericarditis).
13. Known allergy to vaccine components or previous receipt of any experimental adenovirus-vector vaccine by the aerosol route.
14. Enrolment in any clinical trial of experimental treatment for COVID infection within 90 days.
15. For participants in the BAL sub-study, any health-related condition for which study bronchoscopy is contraindicated.
16. For participants in the BAL sub-study, current use of anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Antigen specific T cell responses in blood. | 2 weeks
  Percentage of cytokine positive T cells in the blood
Antigen specific T cell responses in bronchoalveolar lavage (BAL). | 4 weeks
  Percentage of cytokine positive T cells in the BAL
Any grade 3, 4, or 5 adverse events that are possibly or probably related to study vaccine. | 24 weeks
  Frequency, incidence and nature of adverse events

SECONDARY OUTCOMES:
Confirmed COVID infection by reverse transcriptase polymerase chain reaction (RT-PCR) | 24 weeks
  Positive RT-PCR test
CD4 and CD8 T cell responses specific for the spike (S1), nucleoprotein (N) and polymerase (POL) SARS-CoV-2 antigens expressed by the vaccine, including those expressing memory T cell markers, in the peripheral blood. | 4 and 8 weeks
  Percentage of cytokine positive T cells in the blood to specific antigens
Neutralizing and total antibody levels in BAL and blood | 2, 4 and 8 weeks
  Anti-receptor binding domain (RBD) IgG and IgA endpoint titre; percent neutralization (surrogate virus neutralization test [sVNT])
Any adverse events, including grade 1 or 2 or where relationship to vaccine/placebo administration or study procedures is judged not related or unlikely. | 24 weeks
  Frequency, incidence and nature of any adverse events
Tissue-resident memory surface marker expression airway T cells | 4 weeks
  Percentage CD103+CD8+ specific cells

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Smaill, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Canadian Center for Vaccinology, Dalhousie University, Halifax, Nova Scotia
  - Health Sciences Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The full protocol and details of laboratory analyses will be published within 6 months of study enrolment. The statistical analysis plan and individual participant data will be made available to qualified researchers on request.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months following enrolment for protocol and statistical analysis plan. Individual participant data available following analysis.
Access Criteria: Full protocol will be published; statistical analysis plan and individual participant data available on request from qualified researchers